CLINICAL TRIAL: NCT04875039
Title: A Randomized Comparison Between Perineural Dexamethasone and Perineural Mixture of Dexamethasone-Dexmedetomidine as Adjuvants for Ultrasound-Guided Infraclavicular Block
Brief Title: Dexametasone Versus Dexametasone Plus Dexmedetomidine in Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OAIC 1091/19
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Analgesia; Pain, Acute; Upper Extremity Injury
Keywords: dexamethasone; dexmedetomidine; nerve block; adjuvants
MeSH Terms: conditions — Agnosia; Acute Pain; Arm Injuries | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: blinded-randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A research assistant (licensed anesthesiologist) will prepare the local anesthetic solutions and will add the study drug following the randomization order. The operator, patient and investigator assessing the block will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineural dexamethasone (Active Comparator): Addition of dexamethasone 2mg to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: Dexamethasone
- Perineural dexamethasone plus dexmedetomidine (Experimental): Addition of dexamethasone plus dexmedetomidine to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: Dexmedetomidine-Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone 2 mg will be added to the local anesthetic used to block the cords of the brachial plexus with an infraclavicular approach.
  Arms: Perineural dexamethasone
Drug: Dexmedetomidine-Dexamethasone — A mixture of dexamethasone 2mg with dexmedetomidine 50mcg will be added to the local anesthetic used to block the cords of the brachial plexus with an infraclavicular approach.
  Arms: Perineural dexamethasone plus dexmedetomidine

SUMMARY:
This study will compare perineural dexamethasone 2mg and perineural mixture of dexamethasone 2mg plus dexmedetomidine 50mcg DX plus DXD as adjuvants to local anesthetics for ultrasound-guided infraclavicular brachial plexus blocks (ICBs). The protocol is designed as a superiority trial and hypothesizes that the mixture of both drugs results in longer block duration. Furthermore, since analgesic and sensory duration can be influenced by the intake of pain medications and surgical trauma to small cutaneous nerves, respectively, motor block duration was selected as the main outcome to better target the action of both adjuvants on the brachial plexus.

DETAILED DESCRIPTION:
With the approval of Ethics Committee of the Hospital Clínico Universidad de Chile, a total of 50 patients undergoing upper extremity surgery (elbow and below) will be recruited. Recruitment will be carried out by an investigator not involved in patient care in the preoperative clinic or during routine preoperative visits.

All ICBs will be supervised by one of the coauthors and conducted preoperatively in an induction room.

After skin disinfection and draping, the ICB will be performed with a previously described technique. In both groups, a proven 90% effective volume of 35 mL of local anesthetic solution will be injected. As LA solution, it will be used a mixture of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL. The injectate will be slowly injected through the block needle.

Patients will be randomized to receive the study drug, either PN 2 mg dexamethasone or a combination of PN 2 mg dexamethasone with 50 ug dexmedetomidine, mixed with the above-mentioned LA solution.

A research assistant (licensed anesthesiologist) will prepare the local anesthetic solutions and will add the study drug following the randomization order. The operator, patient and investigator assessing the block will be blinded to group allocation.

The primary outcome will be the duration of the motor block (defined as the temporal interval between the end of LA injection through the block needle and the return of movement to the hand and fingers) for patients with successful ICBs. Patients will be provided with a data sheet and asked to record the time at which motor function returns. An investigator blinded to group allocation will collect this data sheet in person (inpatients) or by phone (outpatients) on postoperative day 1.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs)
* Pregnancy
* Prior surgery in the infraclavicular region
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Motor block duration | 24-48 hours after block
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of return of hand and fingers movement

SECONDARY OUTCOMES:
Sensory block duration | Time Frame: 24-48 hours after nerve block
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of the return of hand and fingers sensation
Analgesic block duration | 24-48 hours after nerve block
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of the first sensation of pain in the surgical area
Block performance time | 1 hour before surgery
  Sum of: 1- the acquisition time of the ultrasonographic image. and 2- the time to perform the block itself (from the skin anesthesia to the end of local anesthetic injection)
Intensity of pain during block procedure | 1 hour before surgery
  Evaluated with the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-points score represents the worst imaginable pain. Patients will be asked to rate their pain verbally with this scale. The blinded assessor will register the score reported.
Block onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 14 points out of a maximum of 16 points. The sensorimotor score is described in outcome 7.
Sensory and motor block score | 30 minutes after the ending time of local anesthetic injection
  The sensorimotor block will be assessed every 5 minutes until 30 minutes after the end of local anesthetic injection using a 16-point composite score evaluating sensory and motor block of musculocutaneous, medium, radial, and ulnar nerves.
  Sensation will be assessed with ice in each nerve territory with a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, the patient can feel touch but not cold; 2= anesthetic block, the patient cannot feel cold or touch.
  The motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
  Successful blocks at 30 minutes correlate with a final score ( sum of all individual sensory and motor scores) of at least 14 points out of 16.
Incidence of complete block | 30 minutes after the ending time of local anesthetic injection
  Percentage of blocks with a minimal sensorimotor composite score of 14 points out of a maximum of 16 points at 30 minutes after the injection
Incidence of surgical anesthesia | 30-60 minutes after the ending time of local anesthetic injection
  Ability to proceed with surgery without the need for intravenous narcotics, general anesthesia, rescue blocks or local anesthesia infiltration by the surgeon
Incidence of nerve block side effects | 0 minutes after skin disinfection to 30 minutes after the nerve block
  Determined by the presence of paresthesia, local anesthetic systemic toxicity, vascular puncture, Horner syndrome or hoarseness after the block.
Respiratory depression | 30 minutes after the nerve block to 2 hours after surgery
  Presence of low respiratory rates (lower than 8 breaths per minute) or persistent oxygen requirements (pulse oximetry lower than 90% without supplementary oxygen).
  The respiratory rate and pulse oximetry are continuously measured intra- and post-operatively (in the post-anesthetic care unit) as a standard of care with a multiparameter monitor. Alarms are set to alert when predetermined levels are reached
Bradycardia | 30 minutes after the nerve block to 2 hours after surgery
  Defined as a heart rate lower than 50 beats per minute. The heart rate is continuously measured intra- and post-operatively (in the post-anesthetic care unit) as a standard of care with a multiparameter monitor. Alarms are set to alert when predetermined levels are reached
Hypotension | 30 minutes after the nerve block to 2 hours after surgery
  Mean arterial pressure lower than 60 mmHg. The blood pressure is measured intra- and post-operatively (in the post-anesthetic care unit) as a standard of care with a multiparameter monitor. Alarms are set to alert when predetermined levels are reached
Postoperative persistent sedation | 2 hours after surgery
  Persistent sedation after surgery using Ramsay sedation scale. The scale has 6 points from 1 to 6. A higher score represents a more sedated patient.
  1= anxious, agitated or restless; 2= co-operative, oriented and tranquil; 3= responds to command only; 4= brisk response to light pain or loud auditory stimulus; 5= sluggish response to light pain or loud auditory stimulus; 6= no response.
Persistent neurologic deficit | 7 days after surgery
  Presence of persistent sensory or motor postoperative deficit. The patients will be contacted by telephone and inquired about any sensory or motor deficit in the operated extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran DQ, Bertini P, Zaouter C, Munoz L, Finlayson RJ. A prospective, randomized comparison between single- and double-injection ultrasound-guided infraclavicular brachial plexus block. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):16-21. doi: 10.1097/AAP.0b013e3181c7717c. PMID 20048654
- [Background] Tran DQ, Dugani S, Dyachenko A, Correa JA, Finlayson RJ. Minimum effective volume of lidocaine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):190-4. doi: 10.1097/AAP.0b013e31820d4266. PMID 21270721
- [Background] Leurcharusmee P, Aliste J, Van Zundert TC, Engsusophon P, Arnuntasupakul V, Tiyaprasertkul W, Tangjitbampenbun A, Ah-Kye S, Finlayson RJ, Tran DQ. A Multicenter Randomized Comparison Between Intravenous and Perineural Dexamethasone for Ultrasound-Guided Infraclavicular Block. Reg Anesth Pain Med. 2016 May-Jun;41(3):328-33. doi: 10.1097/AAP.0000000000000386. PMID 27015546
- [Background] Chong MA, Berbenetz NM, Lin C, Singh S. Perineural Versus Intravenous Dexamethasone as an Adjuvant for Peripheral Nerve Blocks: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2017 May/Jun;42(3):319-326. doi: 10.1097/AAP.0000000000000571. PMID 28252523
- [Background] Vorobeichik L, Brull R, Abdallah FW. Evidence basis for using perineural dexmedetomidine to enhance the quality of brachial plexus nerve blocks: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2017 Feb;118(2):167-181. doi: 10.1093/bja/aew411. PMID 28100520
- [Background] Bravo D, Aliste J, Layera S, Fernandez D, Leurcharusmee P, Samerchua A, Tangjitbampenbun A, Watanitanon A, Arnuntasupakul V, Tunprasit C, Gordon A, Finlayson RJ, Tran DQ. A multicenter, randomized comparison between 2, 5, and 8 mg of perineural dexamethasone for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2019 Jan;44(1):46-51. doi: 10.1136/rapm-2018-000032. PMID 30640652
- [Background] Aliste J, Layera S, Bravo D, Fernandez D, Jara A, Garcia A, Finlayson RJ, Tran DQ. Randomized comparison between perineural dexamethasone and dexmedetomidine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2019 Jul 11:rapm-2019-100680. doi: 10.1136/rapm-2019-100680. Online ahead of print. PMID 31300595
- [Derived] Aliste J, Layera S, Bravo D, Aguilera G, Erpel H, Garcia A, Lizama M, Finlayson RJ, Tran D. Randomized comparison between perineural dexamethasone and combined perineural dexamethasone-dexmedetomidine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2022 Jun 21:rapm-2022-103760. doi: 10.1136/rapm-2022-103760. Online ahead of print. PMID 35728840